CLINICAL TRIAL: NCT00325923
Title: A Patient Decision Aid Regarding Natural Health Products for Menopausal Symptoms:a Randomized Controlled Trial
Brief Title: Impact of a Decision Aid Regarding Natural Health Products for Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Laval University (Other); Ottawa Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5-06-03-01
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2006-04

CONDITIONS: Decision Making; Choice Behavior; Decision Support Techniques; Decision Aids
Keywords: Decision making; Decision support; Decisional conflict; Menopause; Natural health products; Herbs; Complementary medicine; Complementary therapies
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Decision aid

SUMMARY:
The aim of this study is to assess the impact of a patient decision aid regarding natural health products for menopausal symptoms on decisional conflict, knowledge and persistence for an option of women aged 45-64 years old. We are expecting a decrease in decisional conflict and an improvement on knowledge level. We are also expecting an intention to use the decision aid in the future and to discuss with the physician or pharmacist about the use, or the intention to use natural health products.

DETAILED DESCRIPTION:
Health decision making is a process known to be difficult, specially in uncertainty context. Because of a lack of evidence, natural health products field remains uncertain. Decision aids (or decision support interventions) have been elaborated in the past for several health decisions and previous studies showed that they seem to be effective on reducing decisional conflict. Following a needs assessment with 40 women and 15 key informants, we developed a decision aid tool specific to the context of natural health products for menopause. In this study, we will assess its impact on decisional conflict, knowledge, persistence for an option, intention to use for a future decision in the same area, and intention to disclose use of natural health products to health professionals.

Comparison: An existing general information brochure on menopause compared to a decision aid tool that we developed based on the Ottawa Decision Support Framework.

ELIGIBILITY:
Inclusion Criteria:

Women :

* between 45 and 64 years old
* reporting suffering from menopausal symptoms
* considering the use of natural health products for menopausal symptoms
* able to read, write, and understand french at a grade 8 level
* able to give an informed consent for her participation to the study

Exclusion Criteria:

* manager and/or owner of a natural health products store,a pharmacy and/or a pharmaceutical company
* person with close relationships with one or many collaborators of this study
* reporting suffering from symptoms with no precise diagnosis

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70
Dates: Start 2006-04; Study Completion 2006-06

PRIMARY OUTCOMES:
Decisional conflict | 2 weeks

SECONDARY OUTCOMES:
Knowledge | 2 weeks
Persistence for an option | 2 weeks
Intention to use for a future decision in the same area | 2 weeks
Intention to disclose use of natural health products to health professionals | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: France Legare, MD, PhD,, Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- Hôpital St-François d'Assise-CHUQ, Québec, Quebec, Canada

REFERENCES:
- [Derived] Legare F, Dodin S, Stacey D, Leblanc A, Tapp S. Patient decision aid on natural health products for menopausal symptoms: randomized controlled trial. Menopause Int. 2008 Sep;14(3):105-10. doi: 10.1258/mi.2008.008014. PMID 18714075